CLINICAL TRIAL: NCT04491825
Title: Diagnostic Classifier for Cutaneous T-cell Lymphomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Patrick M. Brunner, Associate Professor, Medical University of Vienna
Other Study IDs: CTCL_Classifier_KLIF
Record Dates: First submitted 2020-07-23; First posted 2020-07-29 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: CTCL/ Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Suction blister fluid and skin biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mycosis fungoides (MF)
  Interventions: Diagnostic Test: Skin suction blistering and skin biopsies
- Eczema (Atopic Dermatitis)
  Interventions: Diagnostic Test: Skin suction blistering and skin biopsies
- Chronic Plaque-Psoriasis
  Interventions: Diagnostic Test: Skin suction blistering and skin biopsies
- Healthy Control Skin
  Interventions: Diagnostic Test: Skin suction blistering and skin biopsies

INTERVENTIONS:
Diagnostic Test: Skin suction blistering and skin biopsies — Skin suction blistering and skin biopsies will be used for the identification of potential proteomic biomarkers that can distinguish MF from eczema, psoriasis and healthy control skin.

SUMMARY:
Primary cutaneous T-cell lymphomas (CTCL) are a form of skin cancer that is derived from immune cells. The most common form of CTCL is mycosis fungoides (MF). While initially confined to the skin, MF may spread to lymph nodes, blood or inner organs, resulting in an overall poor prognosis for the patient. Thus, being a potentially lethal disease, an early and correct diagnosis of MF has very important implications for the patient. However, diagnosis of early MF is often difficult, as it usually shows a close resemblance to benign inflammatory conditions such as eczema and psoriasis. Strikingly, it takes an average of 3-6 (!) years from the appearance of the first skin lesions until a diagnosis of MF can be made. For this reason, a test to distinguishing early MF from benign inflammatory conditions is urgently mandated. By using skin suction blister fluid as well as skin biopsies from patients with MF, eczema and psoriasis, the investigators want to develop a classifier system that can distinguish early MF from benign inflammatory skin diseases.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and/or histopathological diagnosis of MF, eczema or psoriasis
* Healthy control subjects without personal history of MF, eczema or psoriasis

Exclusion Criteria:

* Ongoing skin-targeted treatment (Wash out times: 2 weeks for topical, and 4 weeks for systemic treatments)
* Ongoing other treatment that might, in the opinion of the investigator, influence proteomic features of the samples to be acquired

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: MF patients need prior histopathological verification of their disease.
  Eczema and psoriasis patients will be diagnosed clinically and, if necessary, on a histopathological basis.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-02-22 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Proteomic signature of MF in comparison to eczema, psoriasis, and healthy control skin | At baseline
  Proteomic multiplex assay

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria